CLINICAL TRIAL: NCT03987321
Title: Retrievability and Incidence of Complex Retrieval in Celect Versus Denali Filter: A Prospective, Randomized, Comparative Study
Brief Title: Retrievability and Incidence of Complex Retrieval in Celect Versus Denali Filter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2019-0020
Record Dates: First submitted 2019-05-26; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Deep Venous Thrombosis
Keywords: Inferior vena cava; filter; deep venous thrombosis; pulmonary embolism; complex retrieval
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Patients who are enrolled in this study are assigned to receive either Denali or Celect filter in the inferior vena cava.
Who Masked: Participant
Masking Description: Participants are blinded to the filter type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denali Group (Experimental): Those who received Denali filter placement
  Interventions: Device: Infrarenal vena cava filter placement
- Celect Group (Experimental): Those who received Celect filter placement
  Interventions: Device: Infrarenal vena cava filter placement

INTERVENTIONS:
Device: Infrarenal vena cava filter placement — Patients who are enrolled in this study are assigned to receive either Denali or Celect filter in the inferior vena cava. All other procedures are the same in both groups

SUMMARY:
The primary purpose of this study is to compare the Celect and Denali filters in terms of complicated filter retrieval and indwelling complications after a 2-month indwelling time.

DETAILED DESCRIPTION:
With anticoagulation being the standard treatment for deep venous thrombosis and pulmonary embolism, inferior vena cava filter placement plays an important role in patients who are amenable to anticoagulant therapy. Currently, many different types of retrievable filters are being used in clinical practice and the choice of the filters depends on operators' preference and institutional availability. Each filter has different designs to maximize retrievability and minimize indwelling complications. Up until now, the prior studies on the filter retrievability and indwelling complications have been retrospective in nature and had relatively long dwell times. Comparative data regarding the retrievability of the inferior vena cava filters may help to choose filter selection. Therefore, the aim of this trial is to compare two commonly used inferior vena cava filters (Denali and Celet filters)

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who develop deep venous thrombosis and/or pulmonary embolism but are good candidates for anticoagulant therapy
* 2. Inferior vena cava filtration before mechanical thrombectomy for deep venous thrombosis
* 3. Prophylactic filter placement because of trauma or major surgery

Exclusion Criteria:

* 1. Sepsis
* 2. Those who need permanent filter placement
* 3. Congenital anatomical anomaly (IVC duplication, interrupted IVC)
* 4. patients who need filter placement in the suprarenal inferior vena cava

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complicated filter retrieval | 2 months after filter placement
  Incidence of retrieval cases that require the use of standard retrieval kit (sheath and snare)

SECONDARY OUTCOMES:
Incidence of penetration | 2 months after filter placement
tilt angle | 2 months after filter placement
Filter migration | 2 months after filter placement
  Filter migration is a change in filter position com-pared with its deployed position (cranial or caudal) of more than 2 cm as documented by diagnostic imaging.
fracture | 2 months after filter placement
  Filter fracture is any loss of a filter's structural integrity(ie, breakage or separation) documented by imaging.
signs of inferior vena cava occlusion/stenosis | 2 months after filter placement
  Any signs of narrowing or obstruction of the IVC where the IVC filter was inserted as documented by CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Severance hospital, Yonsei College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No